CLINICAL TRIAL: NCT05363137
Title: Herramienta De Procesamiento De Lenguaje Natural En Dispositivo Móvil Inteligente Para Fomentar La Adherencia a La Rehabilitación Domiciliaria
Brief Title: Effectiveness of Using a Chatbot to Promote Adherence to Home Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Jose María Blasco Igual, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NLP-PTAdherence
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: Chatbot Assistant
- Control (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Chatbot Assistant — The physiotherpy treatment will be supervised via chatbot
  Arms: Experimental
Other: Standard care — The physiotherpy treatment will be standard care
  Arms: Control

SUMMARY:
A Chatbot oriented to virtually assist patients in a physiotherapy treatment has been designed and developed to interact with patients with musculoskeletal disorders in need for domiciliary rehabilitation. The tool has been designed to promote adherence to rehabilitation, what in turn may have an impact on clinical outcome. A randomized clinical trial involving patients undergoing total knee replacement has bee designed to determine the applicability of the proposal. The participants will be assigned into exerimental group (intervention with the software tool) or control group (standard care).

ELIGIBILITY:
Inclusion Criteria:

* Individuals on the waiting list for total knee replacement surgery
* Undergoing primary total knee replacement surgery
* Who have a personal smartphone
* Who have an instant messaging application installed
* Familiar with the use of such application (more than 3 accesses per week),

Exclusion Criteria:

* Evident cognitive state that prevents to understand care provider instructions
* Vestibular or central nervous system affection (e.g. stroke)
* Cannot read or write
* Do not understand Spanish language
* Not able to consent to participate

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Adherence | Change from baseline to 3 months after surgery date
  Compliance with intervention measured as the percentage of sessions carried out with respect to the total planned

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from baseline to 3 months and one year after surgery date
  Self-administered questionnaire consisting of 24 items divided into pain, stiffness and physical function will register self-reported status. The score is given from 0 to 100
Knee Pain | Change from baseline to 3 months and one year after surgery date
  Measured with a visual analogue scale of pain, being 0 no pain and 10 the worst possible pain

OTHER OUTCOMES:
Safety | Baseline (surgery day) to 12 months
  Adverse events, defined as any unfavorable or unintended diagnosis, sign, symptom, or disease associated with the study
Feasibility_1 | Time from initial day to last day of recruitment up to two years
  Recruitment rate, obtained by dividing the number of participants divided by the number patients invited
Feasibility_2 | Time from initial day to 3 months after surgery date
  Retention rate, obtained by dividing the number of participants assessed at three months by the total number of participants
International Physical Activity Questionnaire (IPAQ-E) | Change from baseline to 3 months after surgery date
  This questionnaire is used to measure the types of intensity of physical activity and sitting time as part of the participants' daily lives, i.e. the total physical activity in MET-min/week and time spent sitting
System Usability | Change from baseline to 3 months after surgery date
  System usability scale will be used for measuring the usability; this consists of a 10 item questionnaire with five response options from Strongly agree to Strongly disagree

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Blasco JM, Diaz-Diaz B, Igual-Camacho C, Perez-Maletzki J, Hernandez-Guilen D, Roig-Casasus S. Effectiveness of using a chatbot to promote adherence to home physiotherapy after total knee replacement, rationale and design of a randomized clinical trial. BMC Musculoskelet Disord. 2023 Jun 15;24(1):491. doi: 10.1186/s12891-023-06607-3. PMID 37322506